CLINICAL TRIAL: NCT01703559
Title: Double-Masked Parallel Evaluation of the Safety and Efficacy of Phentolamine Mesylate Ophthalmic Solution in Subjects With Severe Night Vision Disturbances
Brief Title: The Safety and Efficacy of Phentolamine Mesylate Ophthalmic Solution in Subjects With Severe Night Vision Disturbances
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP-NYX-01a2
Record Dates: First submitted 2012-05-18; First posted 2012-10-10 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Night Vision Complaints; Decrease in Night Vision; Disturbance; Vision, Loss
Keywords: Glare; Starbursts; Halos; Reduced Contrast Sensitivity; Night Vision Disturbances; NVD; NVDs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Administered once daily in both eyes for 15 days
  Interventions: Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo)
- Phentolamine Mesylate Ophthalmic Solution 0.5% (Experimental): Administered once daily in both eyes for 15 days
  Interventions: Drug: Phentolamine Mesylate Ophthalmic Solution 0.5%
- Phentolamine Mesylate Ophthalmic Solution 1.0% (Experimental): Administered once daily in both eyes for 15 days
  Interventions: Drug: Phentolamine Mesylate Ophthalmic Solution 1.0%

INTERVENTIONS:
Drug: Phentolamine Mesylate Ophthalmic Solution 1.0% — Phentolamine mesylate (Nyxol) ophthalmic solution 1.0% is a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol®; Nyxol
  Arms: Phentolamine Mesylate Ophthalmic Solution 1.0%
Drug: Phentolamine Mesylate Ophthalmic Solution 0.5% — Phentolamine mesylate (Nyxol) ophthalmic solution 0.5% is a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol®; Nyxol
  Arms: Phentolamine Mesylate Ophthalmic Solution 0.5%
Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo) — Placebo (vehicle) is a sterile, isotonic, buffered aqueous solution containing mannitol and sodium acetate
  Arms: Placebo

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of phentolamine mesylate 0.5% and 1.0% ophthalmic solution (Nyxol) in the treatment of night vision complaints, including reduced contrast sensitivity
* To evaluate the ocular and systemic safety of phentolamine mesylate 0.5% and 1.0% ophthalmic solution (Nyxol) compared to its vehicle, a sterile, isotonic, buffered aqueous solution containing mannitol and sodium acetate

DETAILED DESCRIPTION:
Randomized, double-masked, multiple dose Phase 2 parallel evaluation of the safety and efficacy of phentolamine mesylate (PM) ophthalmic solution in 60 subjects with severe night vision complaints, evaluating ocular and systemic safety and efficacy following administration of phentolamine mesylate (.05% or 1%) in both eyes for 15 days.

Subjects were randomized into three groups with a 1:1:1 randomization. The groups received either (1) phentolamine mesylate ophthalmic solution 0.5%, (2) phentolamine mesylate ophthalmic solution 1.0%, or (3) placebo, once daily (QD) for 15 days. The treatment period was 15 days, plus 6 additional days over the next 14 days. After 15 days, all subjects were given the opportunity to receive an additional 6 doses of 1.0% phentolamine mesylate to be taken once daily as needed over the next two weeks. There was a post-dosing follow-up evaluation 7 days after the last dose. Study participants completed a night vision questionnaire at pre-treatment and after 15 and 29 days.

Efficacy evaluations included contrast sensitivity (mesopic, with and without glare), mesopic distance high contrast visual acuity (HCVA) and mesopic distance low contrast visual acuity (LCVA). Safety evaluations included photopic distance HCVA, a complete ophthalmic examination and measurement of heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years of age experiencing severe night vision difficulty (as reported subjectively)
2. 0.3 log improvement at least 1 eye using the Holladay Automated Contrast Sensitivity System (HACSS™) test at 2 of 4 spatial frequencies (3, 6, 12, and 18 cycles per degree) under low and high mesopic room illumination with glare
3. Photopic visual acuity (corrected or uncorrected) of 20/25 or better
4. Able and willing to give informed consent and comply with all protocol-mandated procedures

Exclusion Criteria:

1. Cataracts (nuclear sclerosis or anterior subcapsular) of 1+ or greater
2. Contact lens wear within 4 weeks of enrollment
3. Ocular trauma within the past 6 months, or ocular surgery or laser treatment within the past 3 months
4. Refractive surgery or cataract surgery in either eye
5. Use of ocular medication within 4 weeks of Visit 1
6. Clinically significant ocular disease (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca, glaucoma, retinal degenerative disease) which might interfere with the study
7. Any abnormality preventing reliable applanation tonometry of either eye
8. Central corneal thickness greater than 600 µ
9. Known hypersensitivity or contraindication to PM, or any component of the formulation, or to topical anesthetics.
10. Contraindications to phentolamine (including history of myocardial infarction, cerebrovascular spasm, cerebrovascular occlusion, coronary insufficiency, angina, or other evidence suggestive of coronary artery disease)
11. Low blood pressure: systolic < 100 mm Hg or diastolic < 60 mm Hg
12. A history of heart rate abnormalities, such as tachycardia or arrhythmias.
13. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular, or endocrine disorders) which might interfere with the study
14. Use of any systemic alpha adrenergic antagonists up to 4 weeks prior to screening or during the study
15. Changes of systemic medication that could have a substantial effect on ocular autonomic pupil tone 4 weeks prior to screening, or anticipated during the study
16. Participation in any investigational study within the past 30 days
17. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is 1 year post-menopausal or 3 months post-surgical sterilization. All females of childbearing potential must have a negative serum pregnancy test result at the screening examination and must not intend to become pregnant during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2012-04-16 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Eyes With ≥ 0.3 Log Increase in Mesopic Contrast Sensitivities for at Least 2 HACSS Frequencies | Days 1, 4, 8, 15, and 32
  Proportion of eyes with an increase ≥ 0.3 log (2 or more patches) in mesopic contrast sensitivity with glare at one or more frequencies at 1.5, 3, 6, 12, and 18 cycles per degree, measured with the HACSS methodology (categorical analysis)

SECONDARY OUTCOMES:
Pupil Diameter - Change from Day 1 Pre-Dose Baseline | Day 1 post-dose and Days 4, 8, and 15
Mesopic Contrast Sensitivity with Glare at 1 or More Frequencies at 1.5, 3, 6, 12, and 18 Cycles Per Degree, Measured with the HACSS Methodology - Change from Day 1 Pre-Dose Baseline | Day 1 post-dose and Days 4, 8, and 15
Mesopic Contrast Sensitivity without Glare at 1 or More Frequencies at 1.5, 3, 6, 12, and 18 Cycles Per Degree, Measured with the HACSS Methodology - Change from Day 1 Pre-Dose Baseline | Day 1 post-dose and Days 4, 8, and 15
Mesopic Distance High Contrast Visual Acuity (HCVA), Measured with Electronic Early Treatment Diabetic Retinopathy Study (eETDRS) Charts - Change from Day 1 Pre-Dose Baseline | Day 1 post-dose and Days 4, 8, and 15
Mesopic Distance Low Contrast Visual Acuity (LCVA), Measured with eETDRS Charts - Change from Day 1 Pre-Dose Baseline | Day 1 post-dose and Days 4, 8, and 15

OTHER OUTCOMES:
Subjective Evaluations of Vision (NEI Vision Function) - Change from Day 15 | Day 32

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Swearingen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No